CLINICAL TRIAL: NCT03514550
Title: Immunomodulatory Effects of Volatile and Total Intravenous Anesthesia for Patients With Renal Cancer
Brief Title: Effects of Anesthesia on Immunity in Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Efremov Sergey, Principal investigator, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Onko1
Record Dates: First submitted 2018-04-13; First posted 2018-05-02 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Surgery; Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Propofol; Sevoflurane; Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total intravenous anesthesia (Experimental): Patients, scheduled for nephrectomy for kidney cancer will receive neuraxial epidural block and propofol for perioperative anesthesia
  Interventions: Drug: Propofol; Procedure: Epidural block
- Volatile anesthesia (Active Comparator): Patients, scheduled for nephrectomy for kidney cancer will receive neuraxial epidural block and sevoflurane for perioperative anesthesia
  Interventions: Drug: Sevoflurane; Procedure: Epidural block

INTERVENTIONS:
Drug: Propofol — Propofol will be used for anesthesia during surgery
  Arms: total intravenous anesthesia
Drug: Sevoflurane — Sevoflurane will be used for anesthesia during surgery
  Arms: Volatile anesthesia
Procedure: Epidural block — Epidural catheterization Th9-Th10, ropivacaine for perioperative analgesia

SUMMARY:
The aim of the study is a comparative study of the cellular immunity response of patients operated on for kidney cancer under total intravenous and inhalational anesthesia.

DETAILED DESCRIPTION:
The severity of perioperative immunosuppression is directly proportional to the degree of surgical stress. A series of experimental and clinical studies indicate a different effect of certain types of anesthesia on immunity. It is believed that surgical stress itself opens an opportunity for the recurrence of oncological diseases precisely due to the immunosuppressive effect. The aim of present pilot clinical study is to test a hypothesis that total intravenous anesthesia as superior to inhalational anesthesia in term of its effects on cell immunity among patients with kidney cancer.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for renal cancer
* Signed informed concent

Exclusion Criteria:

* Propofol or sevoflurane intolerance
* Contraindications for epidural anesthesia
* Renal failure
* Hepatic failure
* Congestive heart failure
* Previous hemotherapy
* Hematological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
CD 16 | postoperative day 1
  NK cells expression of CD16 receptor

SECONDARY OUTCOMES:
CD45 | Baseline, end of surgery, postoperative days 1, 3-4, 7
  CD45 expression on lymphocytes measured with flow cytometry
CD3 | Baseline, end of surgery, postoperative days 1, 3-4, 7
  CD3 expression on lymphocytes measured with flow cytometry
CD19 | Baseline, end of surgery, postoperative days 1, 3-4, 7
  CD19 expression on lymphocytes measured with flow cytometry
CD4 | Baseline, end of surgery, postoperative days 1, 3-4, 7
  CD4 expression on lymphocytes measured with flow cytometry
CD8 | Baseline, end of surgery, postoperative days 1, 3-4, 7
  CD8 expression on lymphocytes measured with flow cytometry
CD16 | Baseline, end of surgery, postoperative days 1, 3-4, 7
  CD16 expression on lymphocytes measured with flow cytometry
CD25 | Baseline, end of surgery, postoperative days 1, 3-4, 7
  CD25 expression on lymphocytes measured with flow cytometry
HLA-DR | Baseline, end of surgery, postoperative days 1, 3-4, 7
  HLA-DR expression on lymphocytes measured with flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided